CLINICAL TRIAL: NCT03076528
Title: An Innovative Virtually Supervised Exercise for Dialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Hamad Medical Corporation (Industry); Qatar National Research Foundation (QNRF), Award # NPRP 7-1595-3-405 (Unknown)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-38522
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Chronic Kidney Failure; Hemodialysis Complication
Keywords: exercise; exergame; hemodialysis; balance
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with game-based exercise (Experimental): Subjects will be receiving sensor-based interactive ankle & foot exercise program (game-based exercise) during hemo-dialysis, approximately 30 minutes, twice per week and for 4 weeks.
  Interventions: Other: Sensor-based interactive exercise (game-based exercise)
- Non-technology foot and ankle exercise program (Active Comparator): Subjects will be receiving non-technology foot and ankle exercise program during hemodialysis, approximately 30 minutes, twice per week and for 4 weeks.
  Interventions: Other: Non-technology foot and ankle exercise program

INTERVENTIONS:
Other: Sensor-based interactive exercise (game-based exercise) — This intervention includes interactive game-based lower extremity training including repetitive ankle movements in multiple directions. Wearable sensors will provide real-time feedback from foot and ankle position and allow perception of motor-errors during each motor-action
  Arms: Intervention with game-based exercise
Other: Non-technology foot and ankle exercise program — Subjects are asked to perform non-technology based foot and ankle exercises, which include plantar flexion and extension.
  Arms: Non-technology foot and ankle exercise program

SUMMARY:
Among patients with diabetes 35% suffer from chronic renal disease and may require dialysis or kidney replacement over time. Furthermore, in diabetics with end stage renal disease (ESRD) that require dialysis, the risk of foot complications and amputation is even more common, expensive, and devastating. Interestingly, even though incidence of foot ulcers in patients with dialysis has been reported to be same as with patients with history of foot ulcers; dialysis patients have significantly higher rate of foot amputation.

The goal of this research is to incorporate an innovative virtually supervised non-weight bearing exercise in patients undergoing dialysis to reduce risk of fall and foot ulceration by enhancing lower extremity blood flow, joint perception and joint mobility.

Diabetic patients on hemodialysis at Hamad Medical Company will be recruited and will be randomized to either intervention (IG) or control (CG) group and followed for 6 months. The intervention group will take part in a 4-week non-weight bearing exercise program twice per week at the hemodialysis clinic under the supervision of a qualified research staff member. This intervention includes interactive game-based exercises including repetitive ankle and foot movements. Wearable sensors will provide real-time visual/auditory feedback from foot and ankle position and allowed perception of motor-errors during each motor-action. The control group will be instructed to complete a supervised foot and ankle exercise without using sensor technology. Changes in balance, gait, and physical activity, incidence of foot problems will be compared pre- and post-intervention. In addition, the incident of falls, foot ulcers, and limb amputation up to 6 months post intervention will be documented. Investigators hypothesize that patients receiving sensor-based exercises will benefit more compared to group receiving conventional non-technology training in terms of improving functional performance and reducing incidence of foot problems, falls, and limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 50 years or older, who are undergoing hemodialysis process
* Patients in diabetes
* Ability to provide consent

Exclusion Criteria:

* Non-ambulatory patients (unable to walk independently a distance of 20m with or without existence)
* Active foot ulcer
* Major foot amputation
* Charcot neuroarthropathy
* Major hearing/vision impaired
* Any patient with changes in psychotropic or sleep medications in the last 6 weeks
* Patients concurrently participating in another exercise training
* Patients with any clinically significant medical or psychiatric condition, or laboratory abnormality

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-06 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Gait Speed change from Baseline to 4 weeks | Baseline and 4 weeks
  walking ability is quantified by gait speed
Balance change from Baseline to 4 weeks quantified by body sway | Baseline and 4 weeks
  Balance is quantified by body sway

SECONDARY OUTCOMES:
Fear of Falling change from Baseline to 4 weeks using Fall Efficacy Scale International (FES-I) questionnaire | Baseline and 4 weeks
  Measuring fear of falling using Fall Efficacy Scale International (FES-I) questionnaire
Depression change from Baseline to 4 weeks using Center of Epidemiologic Depression Scale (CES-D) questionnaire | Baseline to 4 weeks
  Measuring depression using Center of Epidemiologic Depression Scale (CES-D) questionnaire
Change of Incident of falls | Baseline and 6 months
Change of Incidents of foot problems | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Coorporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified data and associated results will be published in peer-review papers or scientific abstracts.

REFERENCES:
- [Result] Zhou H, Al-Ali F, Rahemi H, Kulkarni N, Hamad A, Ibrahim R, Talal TK, Najafi B. Hemodialysis Impact on Motor Function beyond Aging and Diabetes-Objectively Assessing Gait and Balance by Wearable Technology. Sensors (Basel). 2018 Nov 14;18(11):3939. doi: 10.3390/s18113939. PMID 30441843